CLINICAL TRIAL: NCT03452150
Title: A Phase I Study of D-0316 in Patients With Advanced Non Small Cell Lung Cancer With Mutation of Epidermal Growth Factor Receptor Tyrosine Kinase
Brief Title: D-0316 First Time in Patients Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XY-101
Record Dates: First submitted 2018-02-13; First posted 2018-03-02 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Advanced Non Small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily oral dose of D-0316 (Experimental)
  Interventions: Drug: D-0316

INTERVENTIONS:
Drug: D-0316 — If initial dosing of D-0316 is tolerated then subsequent cohorts will test increasing doses until a maximum tolerated dose or maximum feasible dose is defined

SUMMARY:
This is a phase 1 open label multicentre study of D-0316 administered orally in patients with advanced NSCLC who have progressed following prior therapy with an EGFR-TKI (Epidermal Growth Factor Receptor tyrosine kinase inhibitor agent). This is the first time this drug has ever been tested in patients, and so it will help to understand safety, tolerability, pharmacokinetics and preliminary anti-tumour activity of ascending doses of D-0316.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses
* Histological or cytological confirmation diagnosis of Non Small Cell Lung Cancer (NSCLC).
* Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI e.g. gefitinib or erlotinib. In addition other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.
* Confirmation that the tumour harbours an EGFR T790M mutation.
* No deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks.
* Evaluable or measurable disease per RECIST v1.1

Exclusion Criteria:

* Treatment with an EGFR TKI (erlotinib or gefitinib) within 14 days of the first dose of study treatment.
* Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from the treatment of advanced NSCLC from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | Day 1 - Day 28
  Incidence of DLTs
Adverse events | Day 1 - Day 28
  Incidence of AEs
Laboratory results | Day 1 - Day 28
  Incidence of laboratory abnormalities
Vital signs | Day 1 - Day 28
  Incidence of vital sign abnormalities
Electrocardiogram | Day 1 - Day 28
  Incidence of ECG abnormalities

SECONDARY OUTCOMES:
Pharmacokinetic: area under the plasma concentration versus time curve (AUC) | Day 1 through 6, Cycle Day 1-Day 15
  AUC: area under the plasma concentration versus time curve for D-0316
Pharmacokinetic: maximum plasma drug concentration (Cmax) | Day 1 through 6, Cycle Day 1-Day 15
  Cmax: maximum plasma drug concentration of D-0316
Pharmacokinetic: Time to reach the Cmax (Tmax) | Day 1 through 6, Cycle Day 1-Day 15
  tmax: Time to reach the Cmax of D-0316
Pharmacokinetic: Apparent terminal half-life (t1/2) | Day 1 through 6, Cycle Day 1-Day 15
  t1/2: apparent terminal half-life of D-0316
Antitumor activity | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Antitumor activity by evaluation of tumor response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Research Site, Changchun, Jilin
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Jian H, Wang K, Cheng Y, Ding L, Wang Y, Shi Z, Zhang L, Wang Y, Lu S. Phase I Trial of a Third Generation EGFR Mutant-Selective Inhibitor (D-0316) in Patients with Advanced Non-Small Cell Lung Cancer. Oncologist. 2022 Mar 11;27(3):163-e213. doi: 10.1093/oncolo/oyab007. PMID 35274722